CLINICAL TRIAL: NCT04291404
Title: A Randomized Controlled Trial of Virtual Reality-based Distraction for Venipuncture-related Distress in Children
Brief Title: Virtual Reality-based Distraction to Reduce Distress in the Pediatric Emergency Department
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00095418
Record Dates: First submitted 2020-02-20; First posted 2020-03-02 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2021-10

CONDITIONS: Children Requiring IV Placement
Keywords: Pain; Distress; Virtual Reality; Distraction Therapy
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (Control) Arm (No Intervention): Standard of care treatment, which may include a combination of the following, at the discretion of the treating team and family: parent/ caregiver support, child life services, healthcare provider support, etc.
- Intervention Arm (Experimental): Addition of distraction via an immersive, interactive VR experience to Standard of Care
  Interventions: Device: Virtual Reality Distraction

INTERVENTIONS:
Device: Virtual Reality Distraction — Distraction therapy using a Virtual Reality (VR) device
  Arms: Intervention Arm

SUMMARY:
Needle procedures, such as intravenous (IV) insertions, are among the most commonly performed procedures for children needing medical care. IV insertions are often a painful and stressful experience for both children and their parents/ caregivers. Pediatric pain and distress that is not adequately treated may lead to a frightened and uncooperative child, repeated IV attempts and overall frustration with care for the family and clinical team.

Distraction therapy is a common psychological strategy which involves engaging children in a cognitive task or activity in order to divert attention away from painful stimuli. Given children's growing enthusiasm for novel technology, the investigators propose that an immersive virtual reality (VR) experience may provide an effective means of distraction for children undergoing IV insertions.

DETAILED DESCRIPTION:
Objectives: The investigators' primary objective is to compare the reduction of distress with the use of distraction (via the VR intervention) versus current standard of care in children aged 6 to 17 years who are undergoing IV placement. The secondary objectives are to compare (a) the reduction of pain; (b) the reduction of fear; (c) the reduction of parental/caregiver anxiety; and (d) parental/caregiver and nurse satisfaction with the procedure in the intervention versus control arms; and (e) to assess the safety of using VR intervention in children aged 6 to17 years who are undergoing IV placement.

Research Plan: The investigators will conduct a randomized controlled trial consisting of a control arm receiving departmental standard of care and an intervention arm which will include the addition of an immersive VR experience to current standard of care. Children 6 to 17 years of age who are undergoing IV insertions in the Stollery Children's Hospital emergency department will be considered for enrollment into the study. Approximately 80 families will be recruited over a one-year period.

Study Intervention and Comparison: The VR intervention will aim to provide distraction by immersing the child in an artificial 3-dimensional environment that will engage them for the duration of the IV procedure. The child will wear a head-mounted display ("VR goggles") that will allow them to explore the virtual world through their own visual perspective in 360-degrees. A small handheld controller (optional) can be used to interact with the virtual environment and change settings. The VR goggles will occlude the patient's view of the treatment room, and a pair of noise-cancelling headphones (optional) can be used to further block out ambient hospital sounds. Together, this will provide the child with a unique vivid experience of being fully immersed or "present" inside the 3D virtual world. The control group will receive departmental standard of care which will include topical anesthetic cream (mandatory) and may include parent/caregiver support, child life services, nursing support, etc (at the discretion of the ED clinical care team and the family). At present, there is no single established distraction therapy or routine that is consistently employed for IV procedures within the study site ED. Thus, for pragmatic and ethical considerations, it is felt that the new study VR intervention should be compared to what is currently already in practice (ie. standard of care). Of note, other forms of technology (e.g. smart phones, tablets) will not be prohibited in the control group, if the family chooses to offer them. Due to ethical and pragmatic considerations, children in both groups must receive topical anesthetic cream for IV placement, as it is known to be effective and considered standard of care within the study hospital.

Study Impact: The use of immersive VR technology has previously shown promise in numerous healthcare settings. However, there is still a need for robust evidence regarding its effectiveness in treating pediatric distress associated with IV procedures, particularly in the emergency department. Results of this randomized controlled trial could inform an evidence-based strategy for the management of pediatric distress, which could be used in settings with and without child life specialists.

ELIGIBILITY:
We will include children presenting to the Stollery Children's Hospital ED, based on the eligibility criteria outlined below:

Inclusion Criteria:

1. child aged 6-17 years
2. requires IV placement
3. will receive topical anesthetic cream for IV placement

Exclusion Criteria:

1. medically unstable (CTAS 1, requires immediate IV insertion)
2. unconscious or not fully alert
3. visual, auditory or cognitive or mental health issues precluding safe interaction with the VR intervention
4. conditions that could be exacerbated by the VR environment (as reported by the family), such as: (i) current symptomatic nausea / vomiting / dizziness / migraine; (ii) history of psychosis / hallucinations / epilepsy
5. presence of an infection / injury which could contaminate the VR intervention equipment (as determined by the healthcare team) including but not limited to: (i) open wounds / infections of the head and neck area; (ii) suspected or confirmed methicillin-resistant Staphylococcus aureus (MRSA) colonization
6. screens positive for 'influenza-like illness' (ILI) as per the current SCH ED screening criteria
7. child or parental language barrier precluding the ability to understand and complete study assessments, in the absence of a native language translator
8. previous enrollment in this study

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 84 (Actual)
Dates: Start 2020-09-28 (Actual); Primary Completion 2022-02-12 (Actual); Study Completion 2022-02-12 (Actual)

PRIMARY OUTCOMES:
Child's total distress score during the IV procedure | During the IV placement procedure
  Two RAs will independently observe a videotape of each child and use the Observational Scale of Behavioral Distress - Revised (OSBD-R) to assess children's response behaviors to pain. (0 = no distress, 23.5 = maximum distress)

SECONDARY OUTCOMES:
Child's pain score during the IV procedure | Immediately after IV placement
  Self reported by child using an 11-point verbal Numerical Rating Scale (vNRS) ranging from 0, which indicates no pain, to 10, which indicates the worst possible pain
Child's Fear | Immediately after IV placement
  Self reported by child using the Children's Fear Scale (CFS). This is a five face scale ranging from 0= not scared at all to 4= most scared possible.
Parental anxiety | Immediately after IV placement
  Parent will fill out the State Trait Anxiety Inventory - State Scale Revised Version (STAI-S, Form Y), a validated and commonly used version of STAI, which has improved psychometric properties. The score ranges from 20 to 80, with 80 indicating maximum anxiety.
Parent/ Caregiver Satisfaction | Immediately following the IV procedure
  Self-reported using a 5-point likert scale, ranging from 1 "Not at all satisfied" to 5 "Very satisfied".
Nurse Satisfaction | Immediately following the IV procedure
  Self-reported using a 5-point likert scale, ranging from 1 "Not at all satisfied" to 5 "Very satisfied".
Child Satisfaction | Immediately following the IV procedure
  For children, we will use a a 5-point likert scale ranging from 1 "Not at all happy" to 5 "Very happy".
Frequency of adverse events related to the study intervention | During the IV procedure
  Determined by assessing the frequency of adverse events post intervention. Nausea will be self-rated by children immediately following the intervention, using the Baxter Retching Faces (BARF) scale. This is a six face scale ranging from 0= no nausea at all to 10= most nausea it is possible to feel.
Child's distress during the IV procedure | Immediately after IV placement
  In addition to assessing child distress via the Observational Scale of Behavioral Distress - Revised (primary outcome), we will also ask children to self-report their distress on an 11-point numerical rating scale ranging from 0 "no distress" to 10 "the most distress you can imagine having". While easy to use and previously employed, this scale has not been validated or compared to the validated Observational Scale of Behavioral Distress - Revised.

CONTACTS AND LOCATIONS:
Overall Officials: Samina Ali, MD, Principal Investigator — University of Alberta
Locations (1):
- Stollery Children's Hospital, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ali S, Hudson S, Rajagopal M, Stinson JN, Gourlay K, Ma K, Candelaria P, Vandermeer B, Felkar B, Schreiner K, Proctor A, Hartling L. A Randomized Controlled Trial of Commercially Available Virtual Reality for Intravenous Cannulation-Related Distress in Children. J Pediatr. 2026 Jan;288:114803. doi: 10.1016/j.jpeds.2025.114803. Epub 2025 Sep 15. PMID 40962105
- [Derived] Ali S, Rajagopal M, Stinson J, Ma K, Vandermeer B, Felkar B, Schreiner K, Proctor A, Plume J, Hartling L. Virtual reality-based distraction for intravenous insertion-related distress in children: a study protocol for a randomised controlled trial. BMJ Open. 2022 Mar 30;12(3):e057892. doi: 10.1136/bmjopen-2021-057892. PMID 35354617